CLINICAL TRIAL: NCT02863354
Title: Intravitreal Aflibercept for Retinal Non-Perfusion in Proliferative Diabetic Retinopathy
Acronym: RECOVERY
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Charles C Wykoff, PhD, MD (Other)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor-Investigator, Charles C Wykoff, PhD, MD, Principal Investigator, Greater Houston Retina Research
Organization: Greater Houston Retina Research (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RECOVERY
Record Dates: First submitted 2016-08-04; First posted 2016-08-11 (Estimated); Results first posted 2021-04-21 (Actual); Last update posted 2021-05-24 (Actual); Status verified 2021-05

CONDITIONS: Proliferative Diabetic Retinopathy
MeSH Terms: interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Q4WKS (Experimental): Aflibercept 2 mg every 4 weeks (defined as every 28 days (+ 7 days) and at least 21 days between injections) through week 48. Following week 48, aflibercept 2 mg every 12 weeks through week 96.
  If NV or PDR are worse per pre-specified criteria at week 60, or at any study visit thereafter, the subject will be treated every 4 weeks through the end of the study.
  Interventions: Drug: Aflibercept
- Q12WKS (Experimental): Aflibercept 2 mg every 12-weeks. Subjects will be followed every 4 weeks through week 12, and can be treated if the pre-specified criteria are met. Starting at week 12 if NV or PDR are stable or improved (as assessed by investigator) the subject will be monitored and treated at a 12-week interval through week 48. If NV or PDR are worse per the pre-specified criteria at week 12, or at any study visit thereafter, the subject will be treated monthly through the end of the study.
  At week 52, aflibercept 2 mg every 4 weeks (defined as 28 days (+ 7 days) and at least 21 days between injections) for subjects with visible retinal non-perfusion. If retinal non-perfusion has completely resolved at week 72, aflibercept every 12 weeks through end of study. For subjects without retinal non-perfusion at week 52, aflibercept 2 mg every 12 weeks through the end of study.
  Interventions: Drug: Aflibercept

INTERVENTIONS:
Drug: Aflibercept — Intravitreal injection
  Other Names: Eylea

SUMMARY:
The RECOVERY trial will assess the safety and tolerability of 2 mg intravitreal aflibercept injections (IAI) given monthly (Q4WK) or every 12 weeks (Q12WK) for the treatment of retinal capillary non-perfusion (RNP) associated with proliferative diabetic retinopathy (PDR).

* Assess the safety and tolerability of IAI for the treatment of proliferative diabetic retinopathy by evaluating the incidence and severity of ocular and systemic adverse events through week 52
* Change in area of retinal capillary non-perfusion, as assessed by central reading center, from baseline through week 52

DETAILED DESCRIPTION:
The investigational product is intravitreal aflibercept injection, which will be supplied by Regeneron Pharmaceuticals, Inc. in sterile vials for intravitreal (IVT) injection. Vials must be used (defined as entered with needle) only once. All drug supplies are to be kept under recommended storage conditions.

The injection volume will be 50μL (0.05 mL) and will be administered to the subjects by IVT injection.

Study eyes will be assigned randomly (1:1 ratio) to one of the following 2 treatment arms:

* Group 1- aflibercept 2 mg every 4 weeks (defined as every 28 days (+ 7 days) and at least 21 days between injections) through week 48. Subjects will have a mandatory Year 1 visit at week 48. Subjects have a mandatory visit at week 52 & will not receive treatment. During the second year of follow-up, subjects will be monitored and treated every 12 weeks (Week 60, 72, 84 and 96) with an end of study visit at week 100. If NV or PDR are worse per the pre-specified criteria at week 60, or at any study visit thereafter, the subject will be treated monthly through the end of the study.
* Group 2 - aflibercept 2 mg every 12-weeks for 48 weeks. Subjects will be followed every 4 weeks through week 12, and can be treated if the pre-specified criteria are met. Starting at week 12 if NV or PDR are stable or improved (as assessed by investigator) the subject will be monitored and treated at a 12-week interval through week 48. If NV or PDR are worse per the pre-specified criteria at week 12, or at any study visit thereafter, the subject will be treated monthly through week 48. At week 52 -

  * For subjects without any retinal non-perfusion, monitoring and treatment will continue at every 12 weeks (Week 60, 72, 84, 96) with an end of study visit at week 100.
  * For subjects with visible retinal non-perfusion, monitoring and treatment will be at a 4-week interval (defined as every 28 days + 7 days and at least 21 days between injections). If retinal non-perfusion has completely resolved at week 72, the subject will be switched back to monitoring and treatment every 12 weeks (Week 72, 84, 96).

Pre-specified criteria (subject must meet at least one criterion, which must be documented with imaging):

1. Increased neovascularization
2. Decrease in BCVA by 5 or more letters due to progressive DME or PDR
3. Worsening central subfield diabetic macular edema causing vision loss, with principal investigator or other delegated investigator confirmation
4. Total area of retinal ischemia increases by 10% as determined by the central reading center

Rescue Treatment At any point throughout the study, for either treatment arm, if PDR progresses despite 3 monthly IAI, a fluorescein angiogram will be performed to evaluate PDR progression. PRP will only be permitted after confirmation of PDR progression with the primary

ELIGIBILITY:
Inclusion Criteria:

1. Type 1 or type 2 diabetes mellitus
2. BCVA ETDRS > 20/400 in the study eye
3. Willing and able to comply with clinic visits and study-related procedures
4. Provide signed informed consent
5. Substantial non perfusion (defined as greater than 20 disc areas), as assessed by the investigator
6. Early PDR, as assessed by the investigator, with no vitreous hemorrhage*

   * Early PDR is defined in which PRP can safely be deferred and vitreous hemorrhage that does not obscure the application of PRP

Exclusion Criteria:

1. Any prior systemic anti-VEGF (anti vascular endothelial growth factor) or IVT anti-VEGF treatment in the study eye,
2. SD-OCT (Spectral Domain Optical Coherence Tomography) central subfield thickness measurement of > 320 µm, in the study eye
3. Evidence of infectious ocular infection, in the study eye, at time of screening
4. History of vitreoretinal surgery in the study eye
5. Any prior Panretinal laser photocoagulation (PRP) in the study eye
6. Current vitreous hemorrhage obscuring retinal imaging in the study eye
7. Cataract surgery in the study eye within 4 weeks of Day 0
8. Uncontrolled blood pressure (defined as > 180/110 mm Hg systolic/diastolic, while seated)
9. Significant renal disease defined as a history of chronic renal failure requiring dialysis or renal transplant
10. Tractional Retinal Detachment threatening the macula in the study eye
11. Corticosteroid treatment (intravitreal or peribulbar) in the study eye within 12 weeks of screening
12. Pregnant or breast-feeding women
13. Sexually active men* or women of childbearing potential who are unwilling to practice adequate contraception during the study. Adequate contraceptive measures include stable use of oral contraceptives or other prescription pharmaceutical contraceptives for 2 or more menstrual cycles prior to screening; intrauterine device (IUD); bilateral tubal ligation; vasectomy; condom plus contraceptive sponge, foam, or jelly, or diaphragm plus contraceptive sponge, foam, or jelly.

    * Contraception is not required for men with documented vasectomy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2019-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles C Wykoff, PhD, MD, Principal Investigator — Retina Consultants Houston
Locations (4):
- United States (4):
  - Retina Consultants of Houston/The Medical Center, Houston, Texas
  - Retina Consultants of Houston/Katy office, Katy, Texas
  - Retina Consultants of Houston, Kingwood, Texas
  - Retina Consultants of Houston, The Woodlands, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kempen JH, O'Colmain BJ, Leske MC, Haffner SM, Klein R, Moss SE, Taylor HR, Hamman RF; Eye Diseases Prevalence Research Group. The prevalence of diabetic retinopathy among adults in the United States. Arch Ophthalmol. 2004 Apr;122(4):552-63. doi: 10.1001/archopht.122.4.552. PMID 15078674
- [Background] Klein R, Klein BE, Moss SE. A population-based study of diabetic retinopathy in insulin-using patients diagnosed before 30 years of age. Diabetes Care. 1985 Sep-Oct;8 Suppl 1:71-6. doi: 10.2337/diacare.8.1.s71. PMID 4053957
- [Background] Preliminary report on effects of photocoagulation therapy. The Diabetic Retinopathy Study Research Group. Am J Ophthalmol. 1976 Apr;81(4):383-96. doi: 10.1016/0002-9394(76)90292-0. PMID 944535
- [Background] Writing Committee for the Diabetic Retinopathy Clinical Research Network; Gross JG, Glassman AR, Jampol LM, Inusah S, Aiello LP, Antoszyk AN, Baker CW, Berger BB, Bressler NM, Browning D, Elman MJ, Ferris FL 3rd, Friedman SM, Marcus DM, Melia M, Stockdale CR, Sun JK, Beck RW. Panretinal Photocoagulation vs Intravitreous Ranibizumab for Proliferative Diabetic Retinopathy: A Randomized Clinical Trial. JAMA. 2015 Nov 24;314(20):2137-2146. doi: 10.1001/jama.2015.15217. PMID 26565927
- [Background] Photocoagulation treatment of proliferative diabetic retinopathy. Clinical application of Diabetic Retinopathy Study (DRS) findings, DRS Report Number 8. The Diabetic Retinopathy Study Research Group. Ophthalmology. 1981 Jul;88(7):583-600. PMID 7196564
- [Background] Early photocoagulation for diabetic retinopathy. ETDRS report number 9. Early Treatment Diabetic Retinopathy Study Research Group. Ophthalmology. 1991 May;98(5 Suppl):766-85. PMID 2062512
- [Background] Ferris F. Early photocoagulation in patients with either type I or type II diabetes. Trans Am Ophthalmol Soc. 1996;94:505-37. PMID 8981711
- [Background] Aiello LP, Avery RL, Arrigg PG, Keyt BA, Jampel HD, Shah ST, Pasquale LR, Thieme H, Iwamoto MA, Park JE, et al. Vascular endothelial growth factor in ocular fluid of patients with diabetic retinopathy and other retinal disorders. N Engl J Med. 1994 Dec 1;331(22):1480-7. doi: 10.1056/NEJM199412013312203. PMID 7526212
- [Background] Ip MS, Domalpally A, Hopkins JJ, Wong P, Ehrlich JS. Long-term effects of ranibizumab on diabetic retinopathy severity and progression. Arch Ophthalmol. 2012 Sep;130(9):1145-52. doi: 10.1001/archophthalmol.2012.1043. PMID 22965590
- [Background] Ip MS, Domalpally A, Sun JK, Ehrlich JS. Long-term effects of therapy with ranibizumab on diabetic retinopathy severity and baseline risk factors for worsening retinopathy. Ophthalmology. 2015 Feb;122(2):367-74. doi: 10.1016/j.ophtha.2014.08.048. Epub 2014 Nov 18. PMID 25439595
- [Background] Brown DM, Schmidt-Erfurth U, Do DV, Holz FG, Boyer DS, Midena E, Heier JS, Terasaki H, Kaiser PK, Marcus DM, Nguyen QD, Jaffe GJ, Slakter JS, Simader C, Soo Y, Schmelter T, Yancopoulos GD, Stahl N, Vitti R, Berliner AJ, Zeitz O, Metzig C, Korobelnik JF. Intravitreal Aflibercept for Diabetic Macular Edema: 100-Week Results From the VISTA and VIVID Studies. Ophthalmology. 2015 Oct;122(10):2044-52. doi: 10.1016/j.ophtha.2015.06.017. Epub 2015 Jul 18. PMID 26198808
- [Background] Campochiaro PA, Wykoff CC, Singer M, Johnson R, Marcus D, Yau L, Sternberg G. Monthly versus as-needed ranibizumab injections in patients with retinal vein occlusion: the SHORE study. Ophthalmology. 2014 Dec;121(12):2432-42. doi: 10.1016/j.ophtha.2014.06.011. Epub 2014 Jul 21. PMID 25060610
- [Background] Heier J. The Effect of Intravitreal Aflibercept on Capillary Non-perfusion in Patients with Proliferative Retinopathy and/or Macular Edema Secondary to Proliferative Diabetic Retinopathy and Central Retinal Venous Occlusive Disease (ANDROID Study). Retina Society, Paris, France. 2015.
- [Derived] Babiuch A, Wykoff CC, Hach J, Srivastava S, Talcott KE, Yu HJ, Nittala M, Sadda S, Ip MS, Le T, Hu M, Reese J, Ehlers JP. Longitudinal panretinal microaneurysm dynamics on ultra-widefield fluorescein angiography in eyes treated with intravitreal aflibercept for proliferative diabetic retinopathy in the recovery study. Br J Ophthalmol. 2021 Aug;105(8):1111-1115. doi: 10.1136/bjophthalmol-2020-316952. Epub 2020 Aug 22. PMID 32829304
- [Derived] Alagorie AR, Nittala MG, Velaga S, Zhou B, Rusakevich AM, Wykoff CC, Sadda SR. Association of Intravitreal Aflibercept With Optical Coherence Tomography Angiography Vessel Density in Patients With Proliferative Diabetic Retinopathy: A Secondary Analysis of a Randomized Clinical Trial. JAMA Ophthalmol. 2020 Aug 1;138(8):851-857. doi: 10.1001/jamaophthalmol.2020.2130. PMID 32584384
- [Derived] Babiuch AS, Wykoff CC, Srivastava SK, Talcott K, Zhou B, Hach J, Hu M, Reese JL, Ehlers JP. RETINAL LEAKAGE INDEX DYNAMICS ON ULTRA-WIDEFIELD FLUORESCEIN ANGIOGRAPHY IN EYES TREATED WITH INTRAVITREAL AFLIBERCEPT FOR PROLIFERATIVE DIABETIC RETINOPATHY IN THE RECOVERY STUDY. Retina. 2020 Nov;40(11):2175-2183. doi: 10.1097/IAE.0000000000002727. PMID 31917731

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Eyes
Groups:
- Q4WKS: Aflibercept 2 mg every 4 weeks (defined as every 28 days (+ 7 days) and at least 21 days between injections) through week 48. Following week 48, aflibercept 2 mg every 12 weeks through week 96.
  If NV or PDR are worse per pre-specified criteria at week 60, or at any study visit thereafter, the subject will be treated every 4 weeks through the end of the study.
  Aflibercept: Intravitreal injection
- Q12WKS: Aflibercept 2 mg every 12-weeks. Subjects will be followed every 4 weeks through week 12, and can be treated if the pre-specified criteria are met. Starting at week 12 if NV or PDR are stable or improved (as assessed by investigator) the subject will be monitored and treated at a 12-week interval through week 48. If NV or PDR are worse per the pre-specified criteria at week 12, or at any study visit thereafter, the subject will be treated monthly through the end of the study.
  At week 52, aflibercept 2 mg every 4 weeks (defined as 28 days (+ 7 days) and at least 21 days between injections) for subjects with visible retinal non-perfusion. If retinal non-perfusion has completely resolved at week 72, aflibercept every 12 weeks through end of study. For subjects without retinal non-perfusion at week 52, aflibercept 2 mg every 12 weeks through the end of study.
  Aflibercept: Intravitreal injection
Period: Year 1
Arm/Group | Q4WKS | Q12WKS
Started | 23; 23 Eyes | 20; 20 Eyes
Completed | 19; 19 Eyes | 18; 18 Eyes
Not Completed | 4; 4 Eyes | 2; 2 Eyes
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Death | 0 | 1
Period: Year 2
Arm/Group | Q4WKS | Q12WKS
Started | 19; 19 Eyes | 18; 18 Eyes
Completed | 17; 17 Eyes | 16; 16 Eyes
Not Completed | 2; 2 Eyes | 2; 2 Eyes
Not completed — Lost to Follow-up | 2 | 2

BASELINE CHARACTERISTICS:
Units Other Than Participants: Eyes
Groups:
- Total: Total of all reporting groups
Arm/Group | Q4WKS | Q12WKS | Total
Number analyzed (Participants) | 23 | 20 | 43
Number analyzed (Eyes) | 20 | 20 | 40
Age, Categorical [Count of Units; unit: Eyes]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 4
  >=65 years | 18 | 18 | 36
Age, Continuous [Mean (Inter-Quartile Range); unit: Years] — Population: 3 subjects enrolled were withdrawn early in the trial and replaced.
  Years
    number analyzed (Participants) | 20 | 20 | 40
    (all) | 47.7 [42 to 53] | 48.3 [42 to 58] | 48 [42 to 57]
Sex: Female, Male [Count of Units; unit: Eyes]
  Female | 11 | 8 | 19
  Male | 9 | 12 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: 3 subjects enrolled were withdrawn early in the trial and replaced.
  Participants
    number analyzed (Participants) | 20 | 20 | 40
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 1 | 1 | 2
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 2 | 8 | 10
    White | 13 | 10 | 23
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 4 | 1 | 5
Region of Enrollment [Number; unit: participants] — Population: 3 subjects enrolled were withdrawn early in the trial and replaced.
  participants
    number analyzed (Participants) | 20 | 20 | 40
    United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-related Adverse Events as Assessed by CTCAE v4.0
Description: • Assess the safety and tolerability of IAI for the treatment of proliferative diabetic retinopathy by evaluating the incidence and severity of ocular and systemic adverse events through week 52 and week 100.
Time Frame: 52 and 100 weeks
Population: 3 participants that were enrolled dropped out before their Week 4 visit and were replaced in the study. Thus, only 40 subjects of the original 43 were followed and analyzed in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Q4WKS | Q12WKS
Number analyzed (Participants) | 20 | 20
Participants
  Week 52 | 0 | 0
  Week 100 | 0 | 0

2. Secondary Outcome: Change in Early Treatment of Diabetic Retinopathy Severity Best Corrected Visual Acuity
Description: Mean change in Early Treatment of Diabetic Retinopathy Study Best Corrected Visual Acuity (ETDRS-BCVA) from baseline to week 52 and week 100.
Time Frame: 52 weeks and 100 weeks
Population: 3 participants that were enrolled dropped out before their Week 4 visit and were replaced in the study. Thus, only 40 subjects of the original 43 were followed and analyzed in the study.
  Number analyzed at Week 52 and Week 100 differs from overall number analyzed due to lost to follow up or deceased participants.
Measure: Mean (95% Confidence Interval); unit: ETDRS letters
Arm/Group | Q4WKS | Q12WKS
Number analyzed (Participants) | 20 | 20
ETDRS letters
  Week 52: number analyzed (Participants) | 19 | 17
  Week 52 | 4.26 [0.76 to 7.76] | 4.53 [1.83 to 7.23]
  Week 100: number analyzed (Participants) | 17 | 16
  Week 100 | 4.06 [-0.91 to 9.03] | 8.88 [4.66 to 13.09]

3. Secondary Outcome: Change in Area of Retinal Capillary Non-perfusion Within the Macula
Description: Change in area of retinal capillary non-perfusion within the macula compared to baseline, as assessed by ultrawide-field fluorescein angiogram from baseline to week 52 and week 100.
Time Frame: 52 weeks and 100 weeks
Population: 3 participants that were enrolled dropped out before their Week 4 visit and were replaced in the study. Thus, only 40 subjects of the original 43 were followed and analyzed in the study.
  Number analyzed at Week 52 and Week 100 differs from overall number analyzed due to inability to analyze images, lost to follow up, or deceased participants.
Measure: Mean (Standard Deviation); unit: mm^2
Arm/Group | Q4WKS | Q12WKS
Number analyzed (Participants) | 20 | 20
mm^2
  Week 52: number analyzed (Participants) | 18 | 18
  Week 52 | 0.048 (0.450) | 0.217 (0.388)
  Week 100: number analyzed (Participants) | 17 | 15
  Week 100 | 2.627 (5.171) | 0.940 (1.156)

4. Secondary Outcome: Change in Area of Retinal Capillary Non-perfusion Outside of the Macula
Description: Change in area of retinal capillary non-perfusion outside of the macula from baseline to week 52 and week 100.
Time Frame: 52 weeks and 100 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mm^2
Arm/Group | Q4WKS | Q12WKS
Number analyzed (Participants) | 20 | 20
mm^2
  Week 52: number analyzed (Participants) | 18 | 18
  Week 52 | 182.467 (202.341) | 240.472 (121.967)
  Week 100: number analyzed (Participants) | 17 | 15
  Week 100 | 342.651 (135.957) | 387.204 (169.233)

5. Secondary Outcome: Percentage of Subjects With Neovascularization Regression
Description: Percentage of subjects with neovascularization regression (reduced area of neovascularization) as measured by the central image reading center from baseline to week 52 and week 100.
Time Frame: 52 Weeks and 100 Weeks
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Q4WKS | Q12WKS
Number analyzed (Participants) | 18 | 18
Participants
  Week 52 | 17 | 18
  Week 100: number analyzed (Participants) | 17 | 15
  Week 100 | 17 | 15

6. Secondary Outcome: Percentage of Subjects With Increased Neovascularization
Description: Percentage of subjects with increased neovascularization from baseline to week 52 and week 100.
Time Frame: 52 Weeks and 100 Weeks
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Q4WKS | Q12WKS
Number analyzed (Participants) | 18 | 18
Participants
  Week 52 | 1 | 0
  Week 100: number analyzed (Participants) | 17 | 15
  Week 100 | 0 | 0

7. Secondary Outcome: Percentage of Subjects Who Develop Vitreous Hemorrhage
Description: Percentage of subjects who develop vitreous hemorrhage from baseline to week 52 and week 100.
Time Frame: 52 Weeks and 100 Weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Q4WKS | Q12WKS
Number analyzed (Participants) | 20 | 20
Participants
  Week 52 | 2 | 1
  Week 100 | 4 | 1

8. Secondary Outcome: Percentage of Subjects Treated With Pan-retinal Photocoagulation or Vitrectomy
Description: Percentage of subjects treated with PRP or vitrectomy for progression of PDR from baseline to week 52 and week 100.
Time Frame: 52 Weeks and 100 Weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Q4WKS | Q12WKS
Number analyzed (Participants) | 20 | 20
Participants
  Week 52 | 0 | 0
  Week 100 | 0 | 0

9. Secondary Outcome: Percentage of Subjects Who Develop Center-involving Diabetic Macular Edema
Description: Percentage of subjects, at week 52 and week 100, who develop center-involving diabetic macular edema who did not have center-involving diabetic macular edema at baseline
Time Frame: 52 Weeks and 100 Weeks
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Q4WKS | Q12WKS
Number analyzed (Participants) | 20 | 20
Participants
  Week 52: number analyzed (Participants) | 18 | 18
  Week 52 | 0 | 0
  Week 100: number analyzed (Participants) | 17 | 15
  Week 100 | 0 | 0

10. Secondary Outcome: Changes in Visual Function Outcomes (Self Reported Visual Function)
Description: Changes in self reported visual function utilizing the National Eye Institute Visual Function Questionnaire-25 (NEI VFQ-25) from baseline to week 52 and week 100. The NEI VFQ is a validated measure of patient-reported visual function measured on a scale from 0 (worst function) to 100 (best function).
Time Frame: 52 weeks and 100 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Q4WKS | Q12WKS
Number analyzed (Participants) | 20 | 20
units on a scale
  Week 52: number analyzed (Participants) | 19 | 18
  Week 52 | 6.27 (17.54) | 2.23 (12.86)
  Week 100: number analyzed (Participants) | 15 | 15
  Week 100 | 8.91 (22.04) | 8.82 (13.33)

11. Secondary Outcome: Mean Change in Central Subfield Thickness
Description: Mean change in central subfield thickness (CST) from baseline to week 52 and week 100
Time Frame: 52 weeks and 100 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: micrometers
Arm/Group | Q4WKS | Q12WKS
Number analyzed (Participants) | 20 | 20
micrometers
  Week 52: number analyzed (Participants) | 18 | 18
  Week 52 | -32.947 (20.961) | -20.813 (26.684)
  Week 100: number analyzed (Participants) | 17 | 15
  Week 100 | -35.059 (27.276) | -23.313 (31.979)

12. Secondary Outcome: Change in Area of Total Retinal Capillary Non-perfusion, as Assessed by the Central Reading Center
Description: Change in area of total retinal capillary non-perfusion, as assessed by the central reading center, at week 52 and week 100 compared to baseline.
Time Frame: 52 weeks and 100 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mm^2
Arm/Group | Q4WKS | Q12WKS
Number analyzed (Participants) | 20 | 20
mm^2
  Week 52: number analyzed (Participants) | 18 | 18
  Week 52 | -11.994 (128.697) | 66.752 (100.546)
  Week 100: number analyzed (Participants) | 17 | 15
  Week 100 | 141.317 (110.523) | 245.694 (132.051)

ADVERSE EVENTS:
Time Frame: 52 weeks and 100 weeks
Description: 3 participants that were enrolled dropped out before their Week 4 visit and were replaced in the study. Thus, only 40 subjects of the original 43 were followed and analyzed in the study.
Arm/Group | Q4WKS | Q12WKS
All-Cause Mortality (participants affected / at risk) | 0/20 | 1/20
Serious Adverse Events (participants affected / at risk) | 2/20 | 2/20
Other Adverse Events (participants affected / at risk) | 9/20 | 8/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Q4WKS (N=20) | Q12WKS (N=20)
Worsening of Coronary Artery Disease (Cardiac disorders) | 1 (1) | 0 (0)
NSTEMI (Cardiac disorders) | 1 (1) | 0 (0)
Exacerbation of CHF (Cardiac disorders) | 1 (1) | 0 (0)
Hyperglycemia (Endocrine disorders) | 1 (1) | 0 (0)
Acute Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1)
Bacteremia (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Q4WKS (N=20) | Q12WKS (N=20)
Worsening Cataract (Eye disorders) | 2 (2) | 4 (4)
Subconjunctival Hemorrhage (Eye disorders) | 4 (4) | 0 (0)
Vitreous Hemorrhage (Eye disorders) | 2 (2) | 1 (1)
Floater (Ear and labyrinth disorders) | 2 (2) | 1 (1)
Photophobia (Eye disorders) | 2 (2) | 0 (0)
Eye Pain (Eye disorders) | 1 (1) | 1 (1)
Eye Irritation (Eye disorders) | 2 (2) | 0 (0)
Foreign body sensation (Eye disorders) | 1 (1) | 0 (0)
Ocular Burning (Eye disorders) | 1 (1) | 0 (0)
Dryness (Eye disorders) | 1 (1) | 0 (0)
Corneal Haze (Eye disorders) | 0 (0) | 1 (1)
Acute Follicular Conjunctivitis (Eye disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2017-10-19): https://cdn.clinicaltrials.gov/large-docs/54/NCT02863354/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-03): https://cdn.clinicaltrials.gov/large-docs/54/NCT02863354/SAP_001.pdf